CLINICAL TRIAL: NCT00178997
Title: Realistic Models of Gastrointestinal Bioelectromagnetism
Acronym: SQUID
Status: Completed | Type: Observational
Sponsor: Alan Bradshaw (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Alan Bradshaw, Research Assistant Professor, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 040014; 5R01DK064775 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Ischemia
Keywords: Blood supply; Mesentery
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Good blood flow: Group without ischemia to the small intestine
- Poor blood flow: Groups that have partial ischemia to their small intestine

SUMMARY:
The purpose of this study is to look at the electrical activity present in healthy and diseased smooth muscle of the intestines; and develop both mathematical and computer models.

DETAILED DESCRIPTION:
The Superconducting QUantum Interference Device (SQUID)is a large cylinder machine located in a large shielded room that measures magnetic activity of the intestines. Subjects will be asked to lie underneath and get recordings of the electrical activity of their intestines. They will also be asked to have a CT scan done. From these two procedures, the mathematical and computer models will be developed to determine the difference between normal bowels and those that do not have adequate blood supply.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects and those with diseased bowel

Exclusion Criteria:

* Subjects with claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-02; Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

PRIMARY OUTCOMES:
To observe a difference in the electrical activity between normal and diseased smooth muscle of the intestines. | 2011

SECONDARY OUTCOMES:
To create both mathematical and computer models of the electrical activity of the intestines. | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Leo Cheng, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt UNiversity Medical Center, Nashville, Tennessee, United States